CLINICAL TRIAL: NCT00145938
Title: A Pilot Study of the Effect of Chronic Administration of Sildenafil on Pulmonary Artery Pressure in Patients With Portopulmonary Hypertension
Brief Title: Sildenafil and Pulmonary Artery Pressure
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to complete study
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12562A
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2006-09

CONDITIONS: Pulmonary Hypertension
Keywords: Portopulmonary hypertension; PTPH; pulmonary hypertension; high blood pressure in the pulmonary arteries
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Sildenafil Citrate

INTERVENTIONS:
Drug: sildenafil

SUMMARY:
The purpose of the study is to see if the administration of sildenafil (Viagra) in patients with portopulmonary hypertension could be a safe and effective treatment.

Portopulmonary hypertension (PTPH) is a special type of pulmonary hypertension. Pulmonary hypertension is high blood pressure in the pulmonary arteries that carry unoxygenated blood from the right ventricle of the heart to the lungs. Pulmonary hypertension results from constriction, or tightening, of the blood vessels that supply blood to the lungs. Consequently, it becomes difficult for blood to pass through the lungs, making it harder for the heart to pump blood forward. This stress on the heart leads to enlargement of the heart and eventually fluid can build up in the liver and tissues, such as in the legs. Affected patients can sometimes notice increasing shortness of breath and dizziness.

There is a growing body of evidence suggesting a potential therapeutic role for this sildenafil in patients with primary pulmonary hypertension. Studies are ongoing regarding this area.

Our hypothesis is that chronic oral sildenafil will successfully reduce pulmonary artery pressures by at least 25% (reduction in mean pulmonary artery pressure) and could be an effective treatment for PTPH, especially in candidates for liver transplantation

Primary Hypothesis To measure the effects of a single dose of sildenafil on pulmonary arterial pressure in patients with PTPH

Secondary Hypothesis To measure the effects of chronic (3 month) treatment with sildenafil on pulmonary arterial pressure, safety, and tolerability in patients with PTPH

DETAILED DESCRIPTION:
This is a single center (only takes place at University of Chicago), open-label (doctor and subject know that the subject is taking the experimental drut), pilot study to evaluate the effects of sildenafil on pulmonary artery pressures in patients with portopulmonary hypertension.

Patients who are diagnosed with PTPH after having routine care right heart catheterization will be asked if they are interested in participating. Approximately ten subjects will be enrolled. Subjects will undergo the following experimental procedures as part of their participation in this study: blood laboratory tests, medical history, physical exam, inhaled nitric oxide test, study drug (sildenafil) administration, and a pill count.

Sildenafil will be given to these patients 3 times a day for a 12 week period to see if the study drug can lower their pulmonary artery pressures by at least 25%.

ELIGIBILITY:
Inclusion Criteria:

Candidates for enrollment in this clinical trial are limited to adult patients diagnosed with severe portopulmonary hypertension (PTPH). Specifically, other causes of pulmonary hypertension (PH) such as left ventricular dysfunction, valvular heart disease, chronic lung disease, chronic thromboembolic disease, chronic hypoxemia, rheumatologic conditions, and significant untreated obstructive sleep apnea will be excluded in the usual fashion in patients with underlying portal hypertension and usually cirrhosis. The diagnosis of pulmonary hypertension will be confirmed by invasive hemodynamic measurements (i.e. right heart catheterization) and severe PH is defined as a mean pulmonary artery pressure (MPAP) >35 mmHg. If evidence of right ventricular (RV) dysfunction is present (RV dilation, reduced RV ejection fraction (EF), or elevated RV end-diastolic pressure (>10 mmHg) and the MPAP is 30-35 mmHg, then the patient may be enrolled.

Study participants will be selected from those patients referred for hemodynamic assessment of pulmonary hypertension, such as potential liver transplant recipients. They must be capable of giving informed consent. The University of Chicago referring physician will be contacted for concurrence of agreement.

Exclusion Criteria:

Patients with pulmonary arterial hypertension, but not portopulmonary hypertension will be excluded. Patients will be excluded from consideration if they do not have severe PTPH, if invasive hemodynamic assessment is contraindicated, or if there are any contraindications to sildenafil. Patients with unstable coronary syndromes or otherwise significant unrevascularized coronary artery disease and myocardial ischemia as determined by cardiac stress testing and/or coronary angiography will also be excluded. Moribund patients will not be considered for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2003-09; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Outcome measurement will consist of comparing baseline to treatment hemodynamics both after a single dose and chronic therapy in terms of absolute response as well as the presence of a "significant response" defined as at least a 25% reduction in mean

CONTACTS AND LOCATIONS:
Overall Officials: Allen Anderson, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States